CLINICAL TRIAL: NCT02139852
Title: The Physiological Effects of Capsaicinoid Ingestion on Human Metabolism and Exercise Performance
Brief Title: Capsaicinoid Ingestion, Human Metabolism and Exercise
Acronym: Phase 1
Status: Withdrawn | Type: Observational
Why Stopped: Project abandoned
Sponsor: University of Prince Edward Island (Other)
Collaborators: OmniActive Health Technologies (Industry)
Responsible Party: Principal Investigator, Dr. Jamie Burr, Assistant Professor, University of Prince Edward Island
Other Study IDs: OAHTCAPX-003-2014
Record Dates: First submitted 2014-05-06; First posted 2014-05-15 (Estimated); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Metabolism
MeSH Terms: interventions — Capsaicin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Capsaicin

SUMMARY:
Capsaicinoids (the active ingredient in hot peppers) have been shown to cause a moderate increase in energy expenditure (50 kcal/day) as well as reductions in appetite, energy intake, and (visceral) adiposity. As such, there is considerable interest in capsaicinoid for weight loss supplements. Of particular interest are the recent findings that free-fatty acids in the blood are elevated 2-2.5hrs post ingestion, yet changes in typical cardiovascular or sympathetic nervous tone indicators (heart rate, blood pressure) were unaffected, suggesting some of the negative consequences of other stimulants may be avoided. At present, however, more in depth investigations of the effects on endothelial function, vascular autonomic tone and inflammation are lacking.

The investigators seek to understand the effect of 3 months capsaicinoid ingestion on alterations in body composition, traditional cardiovascular risk factors and cardiovascular function

Hypotheses:

1) Continued use of capsaicinoids will alter resting metabolism substrate use, which will result in moderate (but clinically meaningful) alterations in body composition manifested as a decrease in adiposity. 2) Blood lipids will be unaffected by capsaicinoid use, as will brachial blood pressure. 3) Levels of systemic inflammation may increase slightly, and this could have an effect on vascular reactivity to hyperemic flow or baseline vascular tone. However, previous research suggests that these alterations will not be manifested in autonomic nervous tone assessed by changes in heart rate variability.

DETAILED DESCRIPTION:
Project abandoned

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be male or female
* 18 yr -45yr and free from any known or suspected chronic conditions.
* General health and suitability to participate in an exercise/health research study will be confirmed through use of the PAR-Q+ screening questionnaire

Exclusion Criteria:

* Any participant who has a positive answer to a screening question will be required to seek physician approval prior to any physical exercise.
* Baseline arrhythmia (tachycardia (>100pbm) and systolic or diastolic hypertension (>140/90 mmHg) will also be reason for exclusion.
* During baseline anthropometric assessment we will confirm that participants all fall within a typical BMI range (20-30 kg/m2) of either "normal" weight or "overweight", but not "underweight" or "obese".
* Persons who take cardiovascular medications, metabolic medications, smoke cigarettes, excessively consume alcohol, are prone to heartburn, or have a previous diagnosis of hyperlipidemia or hyperinsulemia will also be excluded

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Project abandoned
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Energy substrate use (Fat vs Carbohydrate contributions to metabolism) | 10 weeks
  Expired gas analysis using a metabolic computer to calculate respiratory exchange rates.

SECONDARY OUTCOMES:
Cardiovascular risk factors | 10 weeks
  Vascular reactivity- endothelial function (Endopat), vascular stiffness (Pulse wave velocity), HRV (heart rate variability), Blood lipid/Glucose panel, blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- UPEI, Charlottetown, Prince Edward Island, Canada